CLINICAL TRIAL: NCT04189211
Title: An Open-Label, Dose Escalation Phase I Clinical Trial on Safety, Tolerability and Pharmacokinetics of BAT8001 for Injection in Patients With HER2-Positive Solid Tumors
Brief Title: A Clinical Trial of BAT8001 on Safety, Tolerability and Pharmacokinetics for Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8001-001-CR
Record Dates: First submitted 2019-11-26; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: HER2-Positive Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1.2mg/kg of BAT8001 (Experimental): BAT8001 100mg/box, 1.2mg/kg IV infusions
  Interventions: Drug: BAT8001
- 2.4mg/kg of BAT8001 (Experimental): BAT8001 100mg/box, 2.4mg/kg IV infusions
  Interventions: Drug: BAT8001
- 3.6mg/kg of BAT8001 (Experimental): BAT8001 100mg/box, 3.6mg/kg IV infusions
  Interventions: Drug: BAT8001
- 4.8mg/kg of BAT8001 (Experimental): BAT8001 100mg/box, 4.8mg/kg IV infusions
  Interventions: Drug: BAT8001
- 6.0mg/kg of BAT8001 (Experimental): BAT8001 100mg/box, 6.0mg/kg IV infusions
  Interventions: Drug: BAT8001

INTERVENTIONS:
Drug: BAT8001 — IV infusions.
  Other Names: Recombinant Humanized Anti-HER2 Monoclonal Antibody-Maytansine Conjugate for Injection

SUMMARY:
An Open-Label, Dose Escalation Phase I Clinical Trial on Safety, Tolerability and Pharmacokinetics of BAT8001 for Injection in Patients with HER2-Positive Solid Tumors (breast cancer or gastric cancer)。

DETAILED DESCRIPTION:
This is an open-label, dose escalation Phase I clinical study in two stages. Stage 1 consists of the first four cycles where the tolerability, safety, pharmacokinetics and immunogenicity of BAT8001 for injections will be studied and preliminary efficacy will be evaluated. Efficacy and safety assessments continue from the fifth cycle until disease progression or intolerable toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced solid tumors refractory to standard treatment or of intolerable or no standard treatment.
2. Patients with breast cancer or gastric cancer (including gastroesophageal junction adenocarcinoma) histopathologically or cytologically diagnosed and tested HER2-positive (IHC 3+ and/or ISH+);
3. At least one measurable lesion according to RECIST version 1.1;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Absence of severe hematopoietic abnormalities, and basically normal heart, lung, liver and kidney functions;
6. Expected survival ≥ 3 months;
7. Left ventricular ejection fraction (LVEF) by ultrasound examinations higher than the lower limit of normal range defined by the study site;
8. The cumulative dose of anthracyclines should meet the following: the cumulative dose must not exceed the equivalent dose of 360 mg/m2 doxorubicin.

Exclusion Criteria:

1. Have active hepatitis B virus or hepatitis C;
2. Patients who are positive for the human immunodeficiency virus;
3. Patients with a history of immunodeficiency, including HIV-positive or other acquired or congenital immunodeficiencies, or a history of organ transplantation;
4. Patients with clinically significant active infection as determined by the investigator;
5. Other concurrent, severe or uncontrollable systemic diseases (such as clinically significant metabolic disorders, poor wound healing, ulcers, etc.);
6. Moderate or severe dyspnea at rest caused by advanced malignant tumors or complications or serious primary lung diseases, or currently requiring continuous oxygen therapy, or currently having interstitial lung disease or pneumonia;
7. Cardiac insufficiency within the past 6 months before enrollment based on the following definitions: Grade ≥ 3 symptomatic congestive heart failure (CHF) according to CTCAE v4.03, or a history of Grade ≥ 2 symptomatic congestive heart failure, transmural myocardial infarction, unstable angina according to New York Heart Association (NYHA) Functional Classification, or severe arrhythmia without proper medicinal control, severe heart block, uncontrolled hypertension, or clinically significant cardiovascular disease;
8. Patients with central nervous system or brain metastasis symptoms, or who have received treatment for central nervous system or brain metastasis within 3 month before the first dose;
9. Grade ≥ 2 peripheral neuropathy ;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | A minimum of 21 days after first dose of BAT8001
  DLT is defined as one of the following as per investigator related to study drug:
  1. Grade ≥ 3 non-hematologic, and non-liver organ toxicities (except for Grade 3 diarrhea, nausea and vomiting in the absence of prophylactics);
  2. Grade ≥ 3 cardiotoxicity, new segmental wall-motion abnormalities, or troponin I ≥ 0.2 ng/mL;
  3. Left ventricular ejection fraction (LVEF) ≤ 45% and a ≥ 10% decrease from baseline;
  4. Grade ≥ 4 thrombocytopenia or anemia;
  5. Grade ≥ 4 t neutropenia that persists for more than 4 days or accompanied by fever > 38.3 °C or persistent fever ≥ 38 °C for more than 1 hour;
  6. Grade ≥ 3 elevation in any one of total bilirubin (TBIL), aspartate transaminase (AST) or alanine transaminase (ALT).
  7. Serum transaminase > 3 × ULN and TBIL > 2 × ULN;
  8. For Grade 2 abnormalities in AST or ALT at baseline, a measurement ≥ 10 × ULN.
Maximum tolerated dosed (MTD) | A minimum of 21 days after first dose of BAT8001
  The highest dose level resulting in a DLT in ≤ 1 of 6 patients was declared the MTD.
Area under the curve (AUC)-BAT8001(antibody-drug conjugate), total antibody and Batansine (a maytansine derivative, which is the 3AA-MDC complex) | pre-infusion (Hour 0), 30 minutes after end of BAT8001 infusion on Day 1 Cycle 1, 2, 3, 4 (each cycle is 21 days) up to approximately 3 months
  AUC will be evaluated and reported for BAT8001 and its metabolites.
Maximum serum drug concentration (Cmax)-BAT8001(antibody-drug conjugate), total antibody and Batansine (a maytansine derivative, which is the 3AA-MDC complex) | pre-infusion (Hour 0), 30 minutes after end of BAT8001 infusion on Day 1 Cycle 1, 2, 3, 4 (each cycle is 21 days) up to approximately 3 months
  Maximum serum concentration (Cmax) immediately after dosing will be evaluated and reported for BAT8001 and its metabolites.
Half-life period(t1/2) | pre-infusion (Hour 0), 30 minutes after end of BAT8001 infusion on Day 1 Cycle 1, 2, 3, 4 (each cycle is 21 days) up to approximately 3 months
  Half-life (t1/2) will be evaluated and reported.
Anti drug antibodies (ADA) | pre-infusion (Hour 0) on Day 1 of Cycle 1, 2, 3, 4 (each cycle is 21 days) up to approximately 3 months
  Plasma level of anti drug antibodies (ADA) correlated with BAT8001 plasma level
Neutralizing anti-drug antibodies (NADA) | pre-infusion (Hour 0) on Day 1 of Cycle 1, 2, 3, 4 (each cycle is 21 days) up to approximately 3 months
  Neutralizing anti-drug antibodies (NADA) correlated with BAT8001

SECONDARY OUTCOMES:
Progression free survival time(PFS) | Baseline to the end of the study (up to 3 years)
  PFS is defined as the time from first dose date until the date of disease progression or death due to any reason, whichever occurs first.
Overall response rate(ORR) | Baseline to the end of the study (up to 3 years)
  determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China